CLINICAL TRIAL: NCT05609643
Title: A Study to Evaluate Safety and Effectiveness of RINVOQ in Adult Participants With Ankylosing Spondylitis in the Real-World Japan (SELECT AXIS RW)
Brief Title: Study to Assess Change in Disease Activity and Adverse Events of RINVOQ in Adult Participants With Ankylosing Spondylitis in the Real-World Japan
Acronym: SELECT AXIS RW
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-963
Record Dates: First submitted 2022-11-07; First posted 2022-11-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; RINVOQ
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rinvoq: Participants will receive Rinvoq as prescribed by their physician according to local label.

SUMMARY:
Axial spondyloarthritis (axSpA), which encompasses radiographic axSpA (r-axSpA, also known as ankylosing spondylitis [AS]) is an immune-mediated inflammatory disease primarily affecting the axial skeleton. This study will assess how effective Rinvoq is in treating axSpA.

Rinvoq is an approved drug for treating axSpA. Approximately 100 adult participants who are prescribed Rinvoq by their physician in accordance with local label will be enrolled in Japan.

Participants will receive Rinvoq as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 52 weeks.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participant with clinical diagnosis of ankylosing spondylitis (AS) and meeting the modified New York Criteria for AS.
* Participant who is administered the first dose of Rinvoq for AS.

Exclusion Criteria:

* Participant with prior treatment by JAK inhibitors.
* Participant currently participating in another clinical study except non-interventional study.
* Participant for whom upadacitinib is contraindicated.
* Participants who are not registered within 14 days after initiation of Rinvoq treatment for AS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult participants with Ankylosing Spondylitis (AS)
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Incidence Percentage of Serious Infection as Adverse Drug Reactions ( ADR) | Up to 52 Weeks
  Incidence of serious drug related adverse reactions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (61):
- Japan (61):
  - Kurotsuchi Orthopaedic Clinic /ID# 251076, Kasugashi, Aichi-ken
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital /ID# 258201, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 254435, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 258204, Toyoake, Aichi-ken
  - Tomita Clinic /ID# 251075, Kashiwa-shi, Chiba
  - Noda Hospital /ID# 254429, Noda, Chiba
  - Yamada Rheumatology Clinic /ID# 264182, Matsuyama, Ehime
  - Matsuyama Red Cross Hospital /ID# 261974, Matsuyama, Ehime
  - Yagi Hospital - Fukuoka /ID# 251078, Fukuoka, Fukuoka
  - Kunou Orthopedic Clinic /ID# 252168, Kitakyushu-shi, Fukuoka
  - Hospital Of The University Of Occupational And Environmental Health, Japan /ID# 252570, Kitakyushu-shi, Fukuoka
  - Zaitsu Orthopedics Clinic /ID# 256998, Onojo-shi, Fukuoka
  - Inoue Hospital /ID# 261959, Takasaki-shi, Gunma
  - National Hospital Organization Asahikawa Medical Center /ID# 268282, Asahikawa, Hokkaido
  - Katayama Orthopedic Rheumatology Clinic /ID# 251071, Asahikawa-shi, Hokkaido
  - Sapporo Rheumatology and immunology clinic /ID# 256175, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 258203, Sapporo, Hokkaido
  - Himeji Medical Center /ID# 255197, Himeji-shi, Hyōgo
  - Kobe Kaisei Hospital /ID# 251073, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 253200, Nishinomiya-shi, Hyōgo
  - Clinic Quest For Rheumatology & Well Being /ID# 268817, Mito, Ibaraki
  - Kanazawa University Hospital /ID# 252170, Kanazawa, Ishikawa-ken
  - Sanuki Municipal Hospital /ID# 251104, Sanuki-shi, Kagawa-ken
  - Kagoshima University Hospital /ID# 256997, Kagoshima, Kagoshima-ken
  - Toranomon Hospital Kajigaya /ID# 260158, Kawasaki-shi, Kanagawa
  - Takahashi Clinic /ID# 252924, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital /ID# 254480, Sagamihara-shi, Kanagawa
  - Sakuragicho Yokohama Clinic /ID# 266671, Yokohama, Kanagawa
  - Yokohama City University Medical Center /ID# 258149, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hosp /ID# 252172, Yokohama, Kanagawa
  - Kyoto Okamoto Memorial Hospital /ID# 255153, Kuse-gun, Kyoto
  - Kyoto University Hospital /ID# 261970, Kyoto, Kyoto
  - Chiyoda Hospital /ID# 251077, Hyuga-shi, Miyazaki
  - National Hospital Organization Miyakonojo Medical Center /ID# 268280, Miyakonojō, Miyazaki
  - University of Miyazaki Hospital /ID# 266669, Miyazaki, Miyazaki
  - Yoshida Internal Medicine Clinic - Sakaki /ID# 268285, Sakaki, Nagano
  - Sasebo Chuo Hospital /ID# 253202, Sasebo-shi, Nagasaki
  - Nagasaki Kita Hospital /ID# 266672, Togitsu, Nagasaki
  - Tenri Hospital /ID# 256996, Tenri-shi, Nara
  - National Hospital Organization Osaka Minami Medical Center /ID# 251072, Kawachinagano Shi, Osaka
  - Kinshukai Infusion Clinic /ID# 251070, Osaka, Osaka
  - Osaka City General Hospital /ID# 258202, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 254436, Osaka, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 260159, Takatsuki-shi, Osaka
  - Koga Community Hospital /ID# 251074, Yaizu, Shizuoka
  - Dokkyo Medical University Hospital /ID# 270947, Mibu, Tochigi
  - Anan Medical Center /ID# 268818, Anan-shi, Tokushima
  - Nishiogu RA Clinic /ID# 266670, Arakawa-ku, Tokyo
  - Juntendo University Hospital /ID# 251103, Bunkyo-ku, Tokyo
  - Institute of Science Tokyo Hospital /ID# 252569, Bunkyo-ku, Tokyo
  - Suzuki Clinic Orthopaedics River City /ID# 254482, Chuo-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center /ID# 270441, Meguro-ku, Tokyo
  - Showa University East Hospital /ID# 267448, Shinagawa, Tokyo
  - Meiyo Immunology & Rheumatology Clinic /ID# 256176, Suginami -ku, Tokyo
  - 500koku Orthopedic Clinic /ID# 268283, Nakaniikawa-gun, Toyama
  - Takaoka Rheumatic Orthopedic Clinic /ID# 252895, Takaoka-shi, Toyama
  - Toyama University Hospital /ID# 251682, Toyama, Toyama
  - Kasugai Clinic /ID# 253201, Fuefuki-shi, Yamanashi
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 252166, Osaka
  - Maeshima Rheumatology Clinic /ID# 251079, Ōita
  - Toyama Hospital /ID# 268281, Toyama

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/